CLINICAL TRIAL: NCT05694390
Title: The Effect of the Use of Sterile Transparent Film Dressing on the Duration of Catheter Stay and the Development of Catheter-Related Complications in Newborns
Brief Title: The Effect of the Use of Sterile Transparent Film Dressing in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Mujde CALIKUSU Incekar, Associate Professor, Yuksek Ihtisas Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YIU-M-CI-004
Record Dates: First submitted 2022-12-22; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Newborn; Peripheral Venous Catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: The group applied sterile transparent film dressing (Experimental): The nurses in the unit were trained by the charge nurse of the clinic on catheter-related complications (infiltration, extravasation, phlebitis, and occlusion), the scales used in the study, and the use of sterile transparent film dressing. In the experimental group, a sterile transparent film dressing was used to fix the catheter and was monitored hourly until the catheter was removed.
  Interventions: Other: Use of sterile transparent film dressing
- Control group: The group applied fixed with a tape (blaster) (No Intervention): The nurses in the unit were trained by the charge nurse of the clinic on catheter-related complications (infiltration, extravasation, phlebitis, and occlusion), the scales used in the study, and the use of sterile transparent film dressing. In the control group, the catheter was fixed with a tape (blaster), routinely used in the clinic, and was monitored hourly until the catheter was removed.

INTERVENTIONS:
Other: Use of sterile transparent film dressing — The nurses in the unit were trained by the charge nurse of the clinic on catheter-related complications (infiltration, extravasation, phlebitis, and occlusion), the scales used in the study, and the use of sterile transparent film dressing. In the experimental group, a sterile transparent film dressing was used to fix the catheter and was monitored hourly until the catheter was removed. The infiltration scale for infants, , the criteria of extravasation (Redness accompanied by a vesicle, tissue necrosis, and ulcer), and The Phlebitis Scale were used to evaluate the catheter site.
  Arms: Experimental group: The group applied sterile transparent film dressing

SUMMARY:
It is important that effective catheter fixation will reduce the risk of catheter unavailability for specific reasons and the incidence of catheter-related complications. The aim of this study was to determine the effect of sterile transparent film dressing and tape methods used in pe- ripheral intravenous catheter application in newborns on the duration of catheter stay and the development of catheter-related complications.

DETAILED DESCRIPTION:
It has been reported that effective catheter fixation will reduce the risk of catheter unavailability for specific reasons and the incidence of catheter-related complications. Intravenous cannulas are usually fixed with a thin board, a bandage, and tape. There is no standard way of using PIVC dressings in Turkey. After the catheter is inserted into the vein, gauze and a blaster, sterile transparent dressing materials, or just a blaster, are used to prevent contact of the fixed part and the area of intervention with the external environment. Transparent dressing used for catheter fixation contribute to a more comfortable evaluation of the catheter entry site. It has been suggested that the use of transparent film dressing may be effective in preventing and early detection of catheter-related complications. Moreover, it was concluded that due to the short duration of the procedure, it reduced the cost of manpower, and nurses could devote more time to other patients.

ELIGIBILITY:
Inclusion Criteria:

* less than 4 kg (due to the infiltration scale criteria)
* PICV was inserted for the first time

Exclusion Criteria:

* existing catheter,
* who has a catheter other than PICV (PICC, umbilical catheter, etc.),
* sterile transparent film dressing, tape, babies with allergies to antiseptic solution and catheter,
* with immunodeficiency, and with skin problems that prevent catheter opening

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The infiltration scale for infants | during catheter removal procedure
  The scale published by the Infusion Nurses Association was revised by Tofani et al. The adaptation of the scale to the newborns was carried out by Calikusu Incekar et al. The scale consists of 5 grades: 0, 1, 2, 3, 4 and is applied to babies under 4 kg. In this study, the infiltration scale was used to determine infiltration and extravasation. In addition to the scale items, the criteria of "Redness accompanied by a vesicle, tissue necrosis, and ulcer" were also considered based on the literature to determine extravasation.
The Phlebitis Scale | during catheter removal procedure
  The phlebitis scale published by the Infusion Nurses Society was used. The scale consists of 5 grades: 0, 1, 2, 3, 4.
Occlusion | during catheter removal procedure
  The nurse checked the infant's catheter site for occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan YILDIZ, PhD, Principal Investigator — Istanbul University - Cerrahpasa; Yağmur GÜL, BSN, Principal Investigator — Istanbul Florence Nightingale Hospital; Ozan UZUNHAN, MD, Principal Investigator — Istanbul Florence Nightingale Hospital
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No